CLINICAL TRIAL: NCT03792568
Title: ALK Inhibitor in Metastatic Colorectal Cancer With ALK Mutation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhan Wang, ALK inhibitor in Metastatuc Colorectal Cancer with ALK mutation., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AICAM
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: ALK mutation; ALK inhibitor; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 1,1'-(4,4'-(((5-chloropyrimidine-2,4-diyl)bis(azanediyl))bis(3-methoxy-4,1-phenylene))bis(piperazine-4,1-diyl))diethanone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALK mutation (Experimental)
  Interventions: Other: ALK Inhibitor

INTERVENTIONS:
Other: ALK Inhibitor — Any ALK inhibitor like crizotinib, alectinib and so on.

SUMMARY:
This clinical trial aims to evaluate the efficacy, safety of ALK inhibitor in Metastatic Colorectal Cancer Patients with ALK mutation.

ELIGIBILITY:
Inclusion Criteria:

Patients should be histologically diagnosed with metastatic colorectal cancer or postoperative recurrence; Patients with ALK mutation(including mutation, fusion, rearrangements ); Patients have measurable lesions; Patients are not available for targeted therapy or patients refuse to receive targeted therapy afer second-line treatment; Over 3 weeks after radiotherapy and the radiotherapy focus was not be measured; Age should be 18-25 years; Performance status should be 0-2; Life expectancy should be more than 12 weeks;

Exclusion Criteria:

Patients underwented major surgery or severe trauma within 4 weeks; Patients allergiced to experimental drugs; Patient ready to give birth or who is pregnant; Patients with brain metastases; Patients with chemotherapy contraindication; Patients could not tolerate chemotherapy; Patients have secondary primary tumor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Respone Rate(ORR) | up to 36months
  Evaluation of tumor burden based on RECIST criteria every 2 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes